CLINICAL TRIAL: NCT01824472
Title: Understanding the Sleep Apnea/Insomnia Interaction: a CPAP/Sham-CPAP Trial
Brief Title: Understanding the Sleep Apnea/Insomnia Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 814153; R34HL109462 (NIH)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CPAP+CC (Active Comparator): Continuous Positive Airway Pressure (CPAP) therapy for sleep apnea and contact control (CC) (placebo/sham for cognitive-behavioral therapy for insomnia)
  Interventions: Device: CPAP; Behavioral: CC
- sham CPAP+CC (Sham Comparator): sham CPAP (ineffective CPAP--placebo/sham for sleep apnea) and contact control (placebo/sham for cognitive-behavioral therapy for insomnia)
  Interventions: Device: sham CPAP; Behavioral: CC
- CPAP+CBT (Active Comparator): CPAP therapy for sleep apnea and cognitive-behavioral therapy (CBT) for insomnia
  Interventions: Device: CPAP; Behavioral: CBT

INTERVENTIONS:
Device: CPAP — Treatment for sleep apnea
  Other Names: Continuous positive airway pressure therapy
  Arms: CPAP+CBT; CPAP+CC
Behavioral: CBT — Treatment for insomnia
  Other Names: Cognitive-Behavioral Therapy for Insomnia
  Arms: CPAP+CBT
Device: sham CPAP — Placebo for sleep apnea
  Other Names: Sham (placebo) continuous positive airway pressure
  Arms: sham CPAP+CC
Behavioral: CC — Placebo (sham) for insomnia
  Other Names: Contact control
  Arms: CPAP+CC; sham CPAP+CC

SUMMARY:
Nearly half of all patients with obstructive sleep apnea have insomnia symptoms, and in some, but not all cases, these insomnia symptoms are caused by the obstructive sleep apnea. The purpose of this study is to find out what type of insomnia symptoms are caused by obstructive sleep apnea and therefore most likely to respond to obstructive sleep apnea treatment with continuous positive airway pressure (also known as CPAP) and if additional treatment with cognitive-behavioral therapy for insomnia is beneficial.

ELIGIBILITY:
Inclusion Criteria:

1. Sleep Apnea
2. Insomnia
3. Age >18

Exclusion Criteria:

1. Sedative/psychoactive drug use recently
2. Other clinically significant sleep disorders
3. Previous treatment for obstructive sleep apnea (OSA)
4. Requires oxygen or bilevel PAP therapy
5. Clinically unstable medical condition
6. Recent shift work
7. Significant alcohol use
8. Other clinically significant causes of insomnia
9. Illicit drug use
10. Prescription stimulants
11. Safety restrictions
12. Unable to treat sleep apnea with positive airway pressure therapy
13. Communication barriers
14. Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CPAP+CC: CPAP therapy for sleep apnea and contact control (placebo/sham for cognitive-behavioral therapy for insomnia)
  CPAP: Treatment for sleep apnea
  CC: Placebo (sham) for insomnia
- CPAP+CBT: CPAP therapy for sleep apnea and cognitive-behavioral therapy for insomnia
  CPAP: Treatment for sleep apnea
  CBT: Treatment for insomnia
Period: Overall Study
Arm/Group | CPAP+CC | Sham CPAP+CC | CPAP+CBT
Started | 17 | 13 | 15
Completed | 16 | 6 | 11
Not Completed | 1 | 7 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 5 | 3
Not completed — Ineligible post randomization&screening | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP+CC | Sham CPAP+CC | CPAP+CBT | Total
Number analyzed (Participants) | 17 | 13 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (11.1) | 49.4 (14.6) | 48.5 (14.6) | 48.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 8 | 22
  Male | 8 | 8 | 7 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 8 | 5 | 22
  White | 5 | 5 | 8 | 18
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1 | 2
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Insomnia Severity Index. Minimum: 0. Maximum: 28. Higher scores mean worse outcome. The outcome measure is reported as a change score in which the score at baseline is subtracted from the score at follow-up, thus the more negative the score, the larger the improvement. The total score represents an addition of the questions totals; there is no specific subscale modification required to calculate the total score.
  units on a scale | 22.4 (3.5) | 22.2 (3.1) | 21.4 (3.0) | 21.9 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index Score
Description: Insomnia Severity Index. Minimum: 0. Maximum: 28. Higher scores mean worse outcome. The outcome measure is reported as a change score in which the score at baseline is subtracted from the score at follow-up, thus the more negative the score, the larger the improvement. The total score represents an addition of the questions totals; there is no specific subscale modification required to calculate the total score.
Time Frame: Between Baseline and Day 42.
Population: Study participants who completed protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CPAP+CC | Sham CPAP+CC | CPAP+CBT
Number analyzed (Participants) | 16 | 6 | 11
score on a scale | -8.2 (6.49) | -7.33 (7.28) | -6.27 (5.9)
Statistical Analysis 1: Comparison: CPAP+CC vs Sham CPAP+CC vs CPAP+CBT; Test type: Superiority; p = 0.8, Kruskal-Wallis; Mean difference compared across 3 groups = 0.43 — Kruskal-Wallis test implemented as "PROC NPAR1WAY" in Statistical Analysis System (SAS v9.4) for a single groupwise comparison. The mean difference (baseline to follow-up) was determined for each group, and this was compared across all 3 groups

ADVERSE EVENTS:
Time Frame: 3 months
Description: We used the clinical trials website definitions
Arm/Group | CPAP+CC | Sham CPAP+CC | CPAP+CBT
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 2/13 | 0/15
Other Adverse Events (participants affected / at risk) | 4/17 | 1/13 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP+CC (N=17) | Sham CPAP+CC (N=13) | CPAP+CBT (N=15)
Kidney problems (Renal and urinary disorders) | 0 | 1 (1) | 0 — Subject was hospitalized for transient kidney problems
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 (2) | 0 — Admitted for diarrhea; resolved and discharged within 1 day. Subject had two episodes, so two serious adverse events reported
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP+CC (N=17) | Sham CPAP+CC (N=13) | CPAP+CBT (N=15)
Atrial Fibrillation (Cardiac disorders) | 0 | 1 (1) | 0 — Recurrent paroxysmal atrial fibrillation
Sinus infection (Infections and infestations) | 1 (1) | 0 | 0 — Sinus infection
Ear ache (Ear and labyrinth disorders) | 1 (1) | 0 | 0 — Ear ache
Mouth pain (General disorders) | 1 (1) | 0 | 0 — Mouth pain
Dizziness (Nervous system disorders) | 0 | 0 | 1 (3) — Dizziness
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 — Neck pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT01824472/Prot_SAP_000.pdf